CLINICAL TRIAL: NCT02287870
Title: Low Epidural Anesthesia With Chloroprocaine Versus Lidocaine: a Prospective, Randomized, Double-blinded Multi-centre Clinical Trial in China
Brief Title: Epidural Anesthesia With Chloroprocaine Versus Lidocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Haibin Dai, Attending Doctor of Department of Anesthesiology, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2007NLY-004
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia
Keywords: Epidural anesthesia; Chloroprocaine; Lidocaine
MeSH Terms: interventions — chloroprocaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroprocaine Group (Experimental): Epidural anesthesia with 3% chloroprocaine.
  Interventions: Drug: Chloroprocaine
- Lidocaine Group (Active Comparator): Epidural anesthesia with 2% lidocaine.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Chloroprocaine — 60 patients undergoing lower limb or lower abdominal surgery from three hospitals in China received 3% chloroprocaine.
  Other Names: Chloroprocaine Hydrochloride
  Arms: Chloroprocaine Group
Drug: Lidocaine — 60 patients undergoing lower limb or lower abdominal surgery from three hospitals in China received 2% lidocaine.
  Other Names: Lidocaine Hydrochloride
  Arms: Lidocaine Group

SUMMARY:
Chinese made chloroprocaine has a rapid onset time, effective methodology, can last for a short time, provides fast motor recovery and causes no significant side effects.

DETAILED DESCRIPTION:
Chloroprocaine hydrochloride is the chloridized local anesthetic of procaine hydrochloride, with twice the anesthetic intensity, four to five times the metabolization and half the side effect of procaine. The chloroprocaine hydrochloride product made in China has been on sale since 2002. To determine the clinical efficacy of low-epidural anesthesia with chloroprocaine versus lidocaine, the investigators carried out a prospective, randomized, double-blinded multi-centre clinical trial. The results demonstrate that epidural anesthesia using chloroprocaine has a more rapid onset time and shorter duration than with lidocaine. It can also provide a reliable sensory and motor block in epidural anesthesia, and is thus a more attractive alternative than lidocaine for middle and short duration surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Weight no more than 80 Kg or not more than 20% of normal weight
* American Society of Anesthesiologists (ASA) grade I or II
* No obstacles in thinking or language communication
* No epidural puncture contraindications such as disturbances of blood coagulation, local infection of the puncture site or use of anticoagulants

Exclusion Criteria:

* Chronic obstructive pulmonary diseases
* Serious heart, liver, renal and metabolic diseases
* Cerebral thrombosis and sequela
* Serious dehydration and electrolyte imbalance
* Neuromuscular diseases
* Pregnant or parturient women
* Abnormal liver and kidney function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Epidural anesthesia effects of chloroprocaine versus lidocaine | Four months (January - April, 2008)
  The effects of epidural anesthesia are assessed by onset time of epidural block, pain free and recovery time, the upper block level and time, the degree of muscle relaxation, and motor recovery time.

SECONDARY OUTCOMES:
Comparison of vital signs between chloroprocaine and lidocaine groups | Four months (January - April, 2008)
  The vital signs are assessed by diastolic blood pressure (DBP), systolic blood pressure (SBP), and pulse oxygen saturation (SpO2).

CONTACTS AND LOCATIONS:
Overall Officials: Weiyan Li, M.D., Study Director — School of Medicine, Nanjing University

REFERENCES:
- [Background] FOLDES FF, McNALL PG. 2-Chloroprocaine: a new local anesthetic agent. Anesthesiology. 1952 May;13(3):287-96. doi: 10.1097/00000542-195205000-00009. No abstract available. PMID 14933832
- [Background] Steinemann TL, Sheikholeslami RR, Klein EF, Prokopius MJ. Short-acting peribulbar anesthesia with 2-chloroprocaine. J Cataract Refract Surg. 2002 Jan;28(1):195-6. doi: 10.1016/s0886-3350(01)00899-9. PMID 11777732
- [Background] Hadzic A, Arliss J, Kerimoglu B, Karaca PE, Yufa M, Claudio RE, Vloka JD, Rosenquist R, Santos AC, Thys DM. A comparison of infraclavicular nerve block versus general anesthesia for hand and wrist day-case surgeries. Anesthesiology. 2004 Jul;101(1):127-32. doi: 10.1097/00000542-200407000-00020. PMID 15220781
- [Background] Liu SS, Ware PD, Rajendran S. Effects of concentration and volume of 2-chloroprocaine on epidural anesthesia in volunteers. Anesthesiology. 1997 Jun;86(6):1288-93; discussion 7A. doi: 10.1097/00000542-199706000-00009. PMID 9197297
- [Background] Sell A, Tein T, Pitkanen M. Spinal 2-chloroprocaine: effective dose for ambulatory surgery. Acta Anaesthesiol Scand. 2008 May;52(5):695-9. doi: 10.1111/j.1399-6576.2008.01639.x. PMID 18419724 (Retraction: PMID 22489994 Acta Anaesthesiol Scand. 2012 May;56(5):667)
- [Result] Marica LS, O'Day T, Janosky JE, Nystrom EU. Chloroprocaine is less painful than lidocaine for skin infiltration anesthesia. Anesth Analg. 2002 Feb;94(2):351-4, table of contents. doi: 10.1097/00000539-200202000-00022. PMID 11812697
- [Result] Marsch SC, Sluga M, Studer W, Barandun J, Scharplatz D, Ummenhofer W. 0.5% versus 1.0% 2-chloroprocaine for intravenous regional anesthesia: a prospective, randomized, double-blind trial. Anesth Analg. 2004 Jun;98(6):1789-1793. doi: 10.1213/01.ANE.0000116929.45557.CE. PMID 15155349
- [Result] Jafari S, Kalstein AI, Nasrullah HM, Hedayatnia M, Yarmush JM, SchianodiCola J. A randomized, prospective, double-blind trial comparing 3% chloroprocaine followed by 0.5% bupivacaine to 2% lidocaine followed by 0.5% bupivacaine for interscalene brachial plexus block. Anesth Analg. 2008 Nov;107(5):1746-50. doi: 10.1213/ane.0b013e318185cd5e. PMID 18931242
- [Result] Bjornestad E, Iversen OL, Raeder J. Similar onset time of 2-chloroprocaine and lidocaine + epinephrine for epidural anesthesia for elective Cesarean section. Acta Anaesthesiol Scand. 2006 Mar;50(3):358-63. doi: 10.1111/j.1399-6576.2006.00937.x. PMID 16480471
- [Result] Casati A, Fanelli G, Danelli G, Berti M, Ghisi D, Brivio M, Putzu M, Barbagallo A. Spinal anesthesia with lidocaine or preservative-free 2-chlorprocaine for outpatient knee arthroscopy: a prospective, randomized, double-blind comparison. Anesth Analg. 2007 Apr;104(4):959-64. doi: 10.1213/01.ane.0000258766.73612.d8. PMID 17377114